CLINICAL TRIAL: NCT04680052
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Tafasitamab Plus Lenalidomide in Addition to Rituximab Versus Lenalidomide in Addition to Rituximab in Patients With Relapsed/Refractory (R/R) Follicular Lymphoma Grade 1 to 3a or R/R Marginal Zone Lymphoma
Brief Title: A Phase 3 Study to Assess Efficacy and Safety of Tafasitamab Plus Lenalidomide and Rituximab Compared to Placebo Plus Lenalidomide and Rituximab in Patients With Relapsed/Refractory (R/R) Follicular Lymphoma or Marginal Zone Lymphoma.
Acronym: InMIND
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCMOR 0208-301; 2023-504684-16-00 (Registry Identifier: EU CT Number); 2020-004407-13 (EudraCT Number)
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Follicular Lymphoma; Marginal Zone Lymphoma
Keywords: MOR00208; INCMOR00208; tafasitamab
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — tafasitamab; Rituximab; Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A : tafasitamab + rituximab + lenalidomide (Experimental): Adult patients with Relapsed/Refractory (R/R) Follicular Lymphoma (FL) Grade 1 to 3a or R/R Marginal Zone Lymphoma (MZL)
  Interventions: Drug: tafasitamab; Drug: rituximab; Drug: lenalidomide
- Arm B : placebo+rituximab+lenalidomide (Placebo Comparator): Adult patients with Relapsed/Refractory (R/R) Follicular Lymphoma (FL) Grade 1 to 3a or R/R Marginal Zone Lymphoma (MZL)
  Interventions: Drug: rituximab; Drug: lenalidomide; Drug: placebo

INTERVENTIONS:
Drug: tafasitamab — tafasitamab will be administered IV for 12 cycles
  Other Names: INCMOR00208; MOR00208
  Arms: Arm A : tafasitamab + rituximab + lenalidomide
Drug: rituximab — Rituximab will be administered IV on cycles 1 - 5
Drug: lenalidomide — Lenalidomide will be administered PO for 12 cycles
Drug: placebo — placebo will be administered IV for 12 cycles
  Arms: Arm B : placebo+rituximab+lenalidomide

SUMMARY:
This is a Phase 3 double-blind, placebo-controlled, randomized study designed to investigate whether tafasitamab and lenalidomide as an add-on to rituximab provides improved clinical benefit compared with lenalidomide as an add-on to rituximab in patients with R/R FL Grade 1 to 3a or R/R MZL.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Grade 1, 2, or 3a FL or nodal MZL, splenic MZL, or extra nodal MZL
* Willingness to avoid pregnancy or fathering children
* In the opinion of the investigator, be able and willing to receive adequate mandatory prophylaxis and/or therapy for thromboembolic events (eg, aspirin 70-325 mg daily or low-molecular-weight heparin)
* Previously treated with at least 1 prior systemic anti-CD20 immunotherapy or chemo-immunotherapy
* Documented relapsed, refractory, or PD after treatment with systemic therapy
* ECOG performance status of 0 to 2

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Any histology other than FL and MZL or clinical evidence of transformed lymphoma
* Prior non-hematologic malignancy
* Congestive heart failure
* HCV positivity, chronic HBV infection or history of HIV infection
* Active systemic infection
* CNS lymphoma involvement
* Any systemic anti-lymphoma and/or investigational therapy within 28 days prior to the start of Cycle 1
* Prior use of lenalidomide in combination with rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2028-08-09 (Estimated)

CONTACTS AND LOCATIONS:
Locations (260):
- United States (38):
  - John Muir Health Clinical Research Center, Concord, California
  - Marin Cancer Care, Greenbrae, California
  - The Oncology Institute of Hope and Innovation, Pasadena, California
  - Sharp Memorial Hospital, San Diego, California
  - Middlesex Hospital Cancer Center, Middletown, Connecticut
  - Smilow Cancer Hospital, New Haven, Connecticut
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Brcr Medical Center, Inc, Plantation, Florida
  - Asclepes Research Centers, Weeki Wachee, Florida
  - Northwest Georgia Oncology Centers,P.C, Marietta, Georgia
  - Straub Medical Center, Honolulu, Hawaii
  - Des Moines Oncology Research Association, Des Moines, Iowa
  - Baptist Health Lexington, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - University of Maryland-Greenebaum Cancer Center, Baltimore, Maryland
  - Cancer Center For Blood Disorders, Bethesda, Maryland
  - Barbara Ann Karmanos Cancer Hospital, Detroit, Michigan
  - Metro-Minnesota Community Oncology Reserch Consortium (Mmcorc), Saint Louis Park, Minnesota
  - Hattiesburg Clinic Hematology, Hattiesburg, Mississippi
  - Roswell Park Cancer Institute, Buffalo, New York
  - Nyu Clinical Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Integris Cancer Institute, Oklahoma City, Oklahoma
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - Prisma Health Upstate, Greenville, South Carolina
  - Prairie Lakes Health Care System, Inc., Watertown, South Dakota
  - Texas Oncology-Baylor Charles A. Sammons, Dallas, Texas
  - The Center For Cancer and Blood Disorders, Fort Worth, Texas
  - Lyndon B Johnson General Hospital, Houston, Texas
  - Md Anderson Cancer Center, Houston, Texas
  - Renovatio Clinical, Spring, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Vista Oncology Inc Ps, Olympia, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington-Seattle Cancer Care Alliance, Seattle, Washington
  - Northwest Medical Specialties Pllc, Tacoma, Washington
- Australia (12):
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Wollongong Hospital - Illawarra Regional Hospital, Wollongong, New South Wales
  - Gold Coast Hospital, Southport, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Northern Hospital, Melbourne, Victoria
  - Western Health, St Albans, Victoria
  - Perth Blood Institute, West Perth, Western Australia
  - Eastern Health, Box Hill
  - Royal Hobart Hospital, Hobart
- Austria (4):
  - Landeskrankenhaus Universitatsklinikum Graz, Graz
  - Innsbruck University Hospital, Innsbruck
  - Kepler Universitat Klinikum, Linz
  - *Krankenhaus*, Vienna
- Belgium (10):
  - Zna Stuivenberg, Antwerp
  - A.Z. St.-Jan-Dienst Hematologie, Bruges
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Ucl Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Dienst Hematologie, Edegem
  - Ghent University Hospital, Ghent
  - Universitair Ziekenhuis (Uz) Leuven, Leuven
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
  - AZ Delta, Roeselare
  - Chu Ucl Namur University Hospital Mont-Godinne, Yvoir
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Queen Elizabeth Ii Health Sciences Centre, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Hospital Maisonneuve Rosemont, Montreal, Quebec
  - McGill University Jewish General Hospital, Montreal, Quebec
  - Chu de Quebec - Universite Laval (Chul), Québec, Quebec
- Czechia (6):
  - University, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Ostrava, Ostrava
  - University Hospital Kralovkse Vinohrady, Prague
  - Vseobecna Fakultni Nemocnice, Prague
  - University Hospital Motol, Prague
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense
  - Sjaellands Universitetshospital Naestved, Roskilde
- Finland (4):
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- France (12):
  - Chu Amiens Picardie - Hopital Sud, Amiens
  - Chu Angers Hotel Dieu Nord, Angers
  - Groupe Bordeaux Nord Aquitaine Gbna Polycliniques - Polyclinique Bordeaux Nord Aquitaine Pbna, Bordeaux
  - Centre Hospitalier Universitaire Chu Dijon Bourgogne - Hopital Francois Mitterrand, Dijon
  - Centre Hospitalier de Versailles - Hopital Andre Mignot, Le Chesnay
  - CHU Nantes, Nantes
  - Hospital Saint-Louis Service Oncologie Medicale, Paris
  - A.P.H. Paris Hopital Cochin, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - Centre Hospitalier de Pontoise, Pontoise
  - Centre Hospitalier Annecy-Genevois, Pringy
  - Chru Hopitaux de Tours Hospital Bretonneau, Tours
- Germany (12):
  - Klinikum St. Marien Amberg, Amberg
  - Klinik Fur Innere Medizin Hamatologie and Onkologie, Berlin
  - Universitatsklinikum Essen, Essen
  - University Clinic Giessen Und Marburg Ukgm, Giessen
  - Universitaetsmedizin Greifswald, Greifswald
  - Statistics and Data Corporation (Sdc), Landshut
  - Universitatsmedizin Der Johannes Gutenberg-Universitat Mainz Iii, Mainz
  - Medizinische Fakultaet Mannheim Der Universitaet Heidelberg, Mannheim
  - Universitatsklinikum Munster, Münster
  - Onkologische Schwerpunktpraxis, Oldenburg
  - Universitarsfrauenklinik Ulm, Ulm
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (4):
  - 251 Air Force General Hospital, Athens
  - General Hospital of Athens Laiko, Athens
  - University Hospital of West Attica - Attikon, Athens
  - University General Hospital of Patras, Pátrai
- Hungary (7):
  - Semmelweis Egyetem, Budapest
  - National Institute of Oncology, Budapest
  - Debreceni Egyetem Klinikai Kozpon Belgyogy Klinika, Debrecen
  - Markhot Ferenc Korhaz, Eger
  - Petz Aladar County Teaching Hospital, Győr
  - Szabolcs-Szatmar-Bereg Megyei Korhazak Es Egyetemi Oktatokorhaz, Nyíregyháza
  - University of Szeged, Szeged
- Ireland (2):
  - Beaumont Hospital, Dublin
  - University Hospital Galway, Galway
- Israel (10):
  - Ha Emek Medical Center, Afula
  - Soroka, Bear Sheva
  - Shamir Medical Center Formerly Assaf Harofeh Medical Center, BEER Yaaqov
  - Wolfson, Holon
  - Shaare Zedek Mc, Jerusalem
  - "Laiko" General Hospital of Athens, Hematology of the First Propaedeutic Internal Medicine Clinic, Jerusalem
  - Hadassah, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - Sheba Medical Center, Tel Litwinsky
- Italy (24):
  - Istituto Tumori Giovanni Paolo Ii Irccs Ospedale Oncologico Bari, Bari
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, Brescia
  - Divisione Clinicizzata Di Ematologia, Brescia
  - Fondazione Del Piemonte Per L Oncologia Ircc Candiolo, Candiolo
  - Divisione Clinicizzata Di Ematologia, Catania
  - Presidio Ospedaliero Vito Fazzi, Lecce
  - Comitato Etico Fondazione Irccs Istituto Nazionale Dei Tumori Milano, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Istituto Nazionale Tumori Irccs Fondazione Pascale, Naples
  - Universita Di Napoli Federico Ii, Napoli
  - Azienda Ospedaliero Universitaria Maggiore Della Carita Di Novara, Novara
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga Orbassano, Orbassano
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia - Cervello, Palermo
  - Fondazione Irccs Policlinico San Matteo, Pavia
  - Ausl Di Placenza Ospedale Guglielmo Da Saliceto, Piacenza
  - Uo Ematologia Univ - Aoup Santa Chiara Pisa, Pisa
  - Ospedale Santa Maria Delle Croci, Ravenna
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Ausl Della Romagna, Rimini
  - Universita Degli Studi Di Roma La Sapienza - Umberto I Policlinico Di Roma - Centro Di Ematologia, Roma
  - Ospedale Sant. Eugenio, Rome
  - Irccs Azienda Ospedaliera Universitaria San Martino, San Martino
  - Azienda Ospedaliero Universitaria Citta Della Salute E Della Scienza, Torino
  - Asugi Ospedale Maggiore, Trieste
- Japan (15):
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Chugoku Center Hospital, Fukuyama-shi
  - Gifu Municipal Hospital, Gifu
  - Kagoshima University Hospital, Kagoshima
  - National Cancer Center Hospital East, Kashiwa-shi
  - Hospital of the University of Occupation and Environmental Health, Kitakyushu-shi
  - Kobe City Medical Center General Hospital, Kobe
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya
  - Iuhw Narita Hospital, Narita
  - Kindai University Hospital, Osakasayama-shi
  - Saitama Medical University Hospital, Saitama
  - Osaka University Hospital, Suita-shi
  - Juntendo University Hospital, Tokyo
  - Mie University Hospital, Tsu
  - Yamagata University Hospital, Yamagata
- Netherlands (5):
  - Amsterdam University Medical Centre, Amsterdam
  - Hospital Rijnstate, Arnhem
  - Medisch Spectrum Twente, Enschede
  - Medisch Centrum Leeuwarden, Leeuwarden
  - HMC, Leidschendam
- Norway (2):
  - Innlandet Hospital Trust, Brumunddal
  - Universitetssykehuset I Trondheim - St. Olavs Hospital, Trondheim
- Poland (10):
  - Szpital Spec Brzozowiepoland, Brzozów
  - Pratia Poznan, Katowice
  - Pratia McM Krakow, Krakow
  - Sp Zoz Szpital Uniwersytecki, Krakow
  - Uniwersytet Medyczny W Lodzi - Klinika Hematologii, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Lublin
  - Specjalistyczny Szpital Onkologiczny, Tomaszów Mazowiecki
  - Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw
  - Institute of Hematology and Transfusion Medicine, Warsaw
  - Uniwersytecki Szpital Kliniczny Im. Jana Mikulicza-Radeckiego, Wroclaw
- Russia (2):
  - Rostov State Medical University, Rostov-on-Don
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
- South Korea (13):
  - Pusan National University Yangsan Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University, Daejeon
  - Gacheon University Gil Medical Center, Incheon
  - Jeonbuk National University Hospital, Jeonju
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Yeoido St.Mary'S Hospital, Seoul
- Spain (26):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital General Unviersitario de Alicante, Alicante
  - Ico Hospital Germans Trias I Pujol, Badalona
  - Hospital Del Mar, Barcelona
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario de Cabuenes, Gijón
  - Institut Catala Doncologia Ico - Hospital Duran I Reynals Location, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Fundacion Jimenez Diaz University Hospital, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Quironsalud Madrid, Madrid
  - Hospital Puerta de Hierro, Majadahonda
  - Hospital Universitario Virgen de La Victoria, Málaga
  - Hospital Universitario Virgen de La Arrixaca, Murcia
  - Hospital Son Llatzer, Palma de Mallorca
  - Consorci Hospitalari Parc Tauli de Sabadell, Sabadell
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio Sevilla, Seville
  - Hospital Universitari Mutua Terrassa, Terrassa
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitari I Politecnic La Fe, Valencia
  - Hospital Universitario de Alava, Vitoria-Gasteiz
- Sweden (3):
  - Karolinska University Hospital Solna, Solna
  - Goetalandsregionen - Uddevalla Sjukhus Us, Uddevalla
  - Uppsala Universitet - Akademiska Sjukhuset, Uppsala
- Switzerland (6):
  - University Hospital of Basel Department of Oncology, Basel
  - Oncological Institute of Southern Switzerland, Bellinzona
  - Inselspital - Universitaetsspital Bern, Bern
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - Universitatsspital Zurich, Zurich
- Taiwan (9):
  - E-Da Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University (Ncku) Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Tri Service General Hospital, Taipei
  - Institutional Review Board Taipei Veterans General Hospital, Taipei
  - Hematology and Medical Oncology Too Foundation Sun Yat Sen Cancer Center, Taipei
- Turkey (Türkiye) (3):
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Ankara University Medical Faculty, Ankara
  - Acibadem Maslak Hospital, Istanbul
- Ukraine (2):
  - Communal Non-Profit Enterprise Regional Center of Oncology, Kharkiv
  - National Cancer Institute of Ministry of Health, Kyiv
- United Kingdom (8):
  - University Hospitals Birmingham Nhs Foundation Trust, Birmingham
  - Bristol Haematology and Oncology Centre, Bristol
  - Leicester Royal Infirmary, Leicester
  - The Royal Marsden Nhs Foundation Trust - Chelsea, London
  - The Christie Nhs Foundation Trust Uk, Manchester
  - James Cook University Hospital, Middlesbrough
  - The Royal Marsden Nhs Foundation Trust - Sutton, Sutton
  - The Royal Wolverhampton Nhs Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- [Derived] Sehn LH, Hubel K, Luminari S, Scholz CW, Salar A, Paneesha S, Wahlin BE, Panayiotidis P, Lee HP, Jimenez-Ubieto A, Sancho JM, Kim TM, Domingo Domenech E, Kumode T, Poh C, Thieblemont C, Deeren D, de Wit E, Arbushites M, Vassallo I, Trneny M; inMIND Study team. Tafasitamab, lenalidomide, and rituximab in relapsed or refractory follicular lymphoma (inMIND): a global, phase 3, randomised controlled trial. Lancet. 2026 Jan 10;407(10524):133-146. doi: 10.1016/S0140-6736(25)01778-7. Epub 2025 Dec 5. PMID 41360064
- See also: A Phase 3 Study to Assess Efficacy and Safety of Tafasitamab Plus Lenalidomide and Rituximab Compared to Placebo Plus Lenalidomide and Rituximab in Patients With Relapsed/ Refractory (R/ R) Follicular Lymphoma or Marginal Zone Lymphoma. — https://incyteclinicaltrials.com/studies/incmor-0208-301

RESULTS

PARTICIPANT FLOW:
Groups:
- FL: Tafasitamab + Rituximab + Lenalidomide: Participants with follicular lymphoma (FL) were randomized to receive tafasitamab 12 milligrams per kilogram (mg/kg) intravenously (IV), administered on Days 1, 8, 15, and 22 of Cycles 1 to 3 and on Days 1 and 15 of Cycles 4 to 12. Participants also received oral lenalidomide (including generics) 20 mg once daily (QD), administered at approximately the same time every day on Days 1 to 21 of Cycles 1 to 12, and rituximab (including biosimilars) 375 mg/meters squared (m^2) IV, administered on Days 1, 8, 15, and 22 of Cycle 1 and on Day 1 of Cycles 2 to 5. A treatment cycle was defined as 28 calendar days.
- FL: Placebo + Rituximab + Lenalidomide: Participants with FL were randomized to receive placebo 0.9% saline solution IV, administered on Days 1, 8, 15, and 22 of Cycles 1 to 3 and on Days 1 and 15 of Cycles 4 to 12. Participants also received oral lenalidomide (including generics) 20 mg QD, administered at approximately the same time every day on Days 1 to 21 of Cycles 1 to 12, and rituximab (including biosimilars) 375 mg/m^2 IV, administered on Days 1, 8, 15, and 22 of Cycle 1 and on Day 1 of Cycles 2 to 5. A treatment cycle was defined as 28 calendar days.
- MZL: Tafasitamab + Rituximab + Lenalidomide: Participants with marginal zone lymphoma (MZL) were randomized to receive tafasitamab 12 mg/kg IV, administered on Days 1, 8, 15, and 22 of Cycles 1 to 3 and on Days 1 and 15 of Cycles 4 to 12. Participants also received oral lenalidomide (including generics) 20 mg QD, administered at approximately the same time every day on Days 1 to 21 of Cycles 1 to 12, and rituximab (including biosimilars) 375 mg/m^2 IV, administered on Days 1, 8, 15, and 22 of Cycle 1 and on Day 1 of Cycles 2 to 5. A treatment cycle was defined as 28 calendar days.
- MZL: Placebo + Rituximab + Lenalidomide: Participants with MZL were randomized to receive placebo 0.9% saline solution IV, administered on Days 1, 8, 15, and 22 of Cycles 1 to 3 and on Days 1 and 15 of Cycles 4 to 12. Participants also received oral lenalidomide (including generics) 20 mg QD, administered at approximately the same time every day on Days 1 to 21 of Cycles 1 to 12, and rituximab (including biosimilars) 375 mg/m^2 IV, administered on Days 1, 8, 15, and 22 of Cycle 1 and on Day 1 of Cycles 2 to 5. A treatment cycle was defined as 28 calendar days.
Period: Overall Study
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Started | 273 | 275 | 53 | 53
Completed | 0 | 0 | 0 | 0
Not Completed | 273 | 275 | 53 | 53
Not completed — Ongoing | 244 | 229 | 39 | 46
Not completed — Death | 15 | 22 | 7 | 1
Not completed — Lost to Follow-up | 3 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 11 | 19 | 7 | 5
Not completed — Missing | 0 | 1 | 0 | 0
Not completed — Hypersensitivity to Rituximab; Did Not Receive Treatment | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide | Total
Number analyzed (Participants) | 273 | 275 | 53 | 53 | 654
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (10.89) | 63.7 (11.69) | 68.3 (10.69) | 67.9 (11.40) | 64.8 (11.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 126 | 27 | 26 | 302
  Male | 150 | 149 | 26 | 27 | 352
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 24 | 4 | 8 | 67
  Not Hispanic or Latino | 228 | 226 | 45 | 41 | 540
  Unknown or Not Reported | 14 | 25 | 4 | 4 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 219 | 219 | 43 | 41 | 522
  Black or African-American | 1 | 0 | 0 | 1 | 2
  Asian | 40 | 42 | 7 | 6 | 95
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Not Reported | 11 | 10 | 3 | 4 | 28
  Captured as "Other" in Database | 2 | 4 | 0 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: FL Population: Progression-free Survival (PFS) by Investigator Assessment, Using the Lugano 2014 Criteria, Defined as the Time From Randomization to the First Documented Disease Progression (PD), or Death From Any Cause, Whichever Occurred First
Description: PD, positron emission tomography (PET): score 4 (uptake moderately > liver) or 5 (uptake markedly higher than liver and/or new lesions) for lymph node/extra lymphatic sites with increase in intensity of Baseline uptake and/or new fluorodeoxyglucose (FDG)-avid foci consistent with lymphoma at interim/end-of-treatment assessment; new/recurrent FDG-avid foci in bone marrow; new FDG-avid foci consistent with lymphoma versus other etiology in new lesions. PD, computed tomography (CT): abnormal individual node/lesion with longest diameter (LDi ) >1.5 centimeters (cm) and increase by ≥50% from the product of the perpendicular diameters (PPD) nadir and increase in LDi or shortest diameter (SDi) from nadir; new/clear progression of preexisting nontarget lesions; new/recurrent splenomegaly and bone marrow involvement; regrowth of previously resolved lesions. New node >1.5 cm in any axis. New extranodal site >1.0 cm in any axis; if <1.0 cm, presence is unequivocal and attributable to lymphoma.
Time Frame: up to approximately 34 months
Population: Follicular Lymphoma (FL) Full Analysis Set: all randomized participants with FL. The 2-sided 95% confidence intervals were calculated using the method of Brookmeyer and Crowley with log-log transformation. Censored participants were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 273 | 275 | 0 | 0
months | 22.37 [19.22 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 13.93 [11.53 to 16.39] |  |

2. Primary Outcome: FL Population: Kaplan-Meier Estimates of PFS by Investigator Assessment, Using the Lugano 2014 Criteria, Defined as the Time From Randomization to the First Documented PD, or Death From Any Cause, Whichever Occurred First
Description: PD, PET: score 4 (uptake moderately > liver) or 5 (uptake markedly higher than liver and/or new lesions) for lymph node/extra lymphatic sites with increase in intensity of Baseline uptake and/or new FDG-avid foci consistent with lymphoma at interim/end-of-treatment assessment; new/recurrent FDG-avid foci in bone marrow; new FDG-avid foci consistent with lymphoma versus other etiology in new lesions. PD, CT: abnormal individual node/lesion with LDi >1.5 cm and increase by ≥50% from the PPD nadir and increase in LDi or SDi from nadir; new/clear progression of preexisting nontarget lesions; new/recurrent splenomegaly and bone marrow involvement; regrowth of previously resolved lesions. New node >1.5 cm in any axis. New extranodal site >1.0 cm in any axis; if <1.0 cm, presence is unequivocal and attributable to lymphoma. Kaplan-Meier estimates indicate the percent probability of a participant being alive at the indicated time after treatment start.
Time Frame: up to 2 years
Population: FL Full Analysis Set. Censored participants were included in the analysis. The number of participants analyzed for the Kaplan-Meier estimate at each time point refers to the total number of participants in the analysis set.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 273 | 275 | 0 | 0
percent probability
  6 months | 92.4 [88.3 to 95.1] | 78.2 [72.7 to 82.7] |  |
  12 months | 79.0 [72.8 to 84.0] | 54.0 [47.1 to 60.5] |  |
  18 months | 61.9 [53.4 to 69.3] | 38.5 [30.8 to 46.1] |  |
  2 years | 41.7 [28.4 to 54.6] | 31.8 [23.6 to 40.2] |  |
Statistical Analysis 1: Comparison: FL: Tafasitamab + Rituximab + Lenalidomide vs FL: Placebo + Rituximab + Lenalidomide; Test type: Superiority; p < 0.0001, stratified Log Rank; Hazard Ratio (HR) = 0.434, 95% CI 2-sided [0.324 to 0.580] — The hazard ratio was estimated using a stratified Cox proportional hazards model

3. Secondary Outcome: Overall Population: PFS by Investigator Assessment, Using the Lugano 2014 Criteria, Defined as the Time From Randomization to the First Documented PD, or Death From Any Cause, Whichever Occurred First
Description: PD, PET: score 4 (uptake moderately > liver) or 5 (uptake markedly higher than liver and/or new lesions) for lymph node/extra lymphatic sites with increase in intensity of Baseline uptake and/or new FDG-avid foci consistent with lymphoma at interim/end-of-treatment assessment; new/recurrent FDG-avid foci in bone marrow; new FDG-avid foci consistent with lymphoma versus other etiology in new lesions. PD, CT: abnormal individual node/lesion with LDi >1.5 cm and increase by ≥50% from the PPD nadir and increase in LDi or SDi from nadir; new/clear progression of preexisting nontarget lesions; new/recurrent splenomegaly and bone marrow involvement; regrowth of previously resolved lesions. New node >1.5 cm in any axis. New extranodal site >1.0 cm in any axis; if <1.0 cm, presence is unequivocal and attributable to lymphoma.
Time Frame: up to approximately 34 months
Population: Overall Full Analysis Set. As pre-specified in the Statistical Analysis Plan, the MZL population was considered as a subpopulation of interest, not a main analysis population. The FL and MZL populations were combined for analysis into the Overall population, which was a main analysis population. The 2-sided 95% confidence intervals were calculated using the method of Brookmeyer and Crowley with log-log transformation. Censored participants were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- FL and MZL: Tafasitamab + Rituximab + Lenalidomide: Participants with FL and MZL were randomized to receive tafasitamab 12 mg/kg IV, administered on Days 1, 8, 15, and 22 of Cycles 1 to 3 and on Days 1 and 15 of Cycles 4 to 12. Participants also received oral lenalidomide (including generics) 20 mg QD, administered at approximately the same time every day on Days 1 to 21 of Cycles 1 to 12, and rituximab (including biosimilars) 375 mg/m^2 IV, administered on Days 1, 8, 15, and 22 of Cycle 1 and on Day 1 of Cycles 2 to 5. A treatment cycle was defined as 28 calendar days.
- FL and MZL: Placebo + Rituximab + Lenalidomide: Participants with FL and MZL were randomized to receive placebo 0.9% saline solution IV, administered on Days 1, 8, 15, and 22 of Cycles 1 to 3 and on Days 1 and 15 of Cycles 4 to 12. Participants also received oral lenalidomide (including generics) 20 mg QD, administered at approximately the same time every day on Days 1 to 21 of Cycles 1 to 12, and rituximab (including biosimilars) 375 mg/m^2 IV, administered on Days 1, 8, 15, and 22 of Cycle 1 and on Day 1 of Cycles 2 to 5. A treatment cycle was defined as 28 calendar days.
Arm/Group | FL and MZL: Tafasitamab + Rituximab + Lenalidomide | FL and MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 326 | 328
months | 23.95 [22.34 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 16.39 [13.86 to 18.66]

4. Secondary Outcome: Overall Population: Kaplan-Meier Estimates of PFS by Investigator Assessment, Using the Lugano 2014 Criteria, Defined as the Time From Randomization to the First Documented PD, or Death From Any Cause, Whichever Occurred First
Description: as for outcome 2
Time Frame: up to 2 years
Population: Overall Full Analysis Set. As pre-specified in the Statistical Analysis Plan, the MZL population was considered as a subpopulation of interest, not a main analysis population. The FL and MZL populations were combined for analysis into the Overall population, which was a main analysis population. Censored participants were included in the analysis. The number of participants analyzed for the Kaplan-Meier estimate at each time point refers to the total number of participants in the analysis set.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | FL and MZL: Tafasitamab + Rituximab + Lenalidomide | FL and MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 326 | 328
percent probability
  6 months | 92.7 [89.0 to 95.1] | 80.0 [75.0 to 84.0]
  12 months | 79.7 [74.1 to 84.2] | 58.7 [52.4 to 64.4]
  18 months | 64.1 [56.7 to 70.6] | 44.7 [37.6 to 51.5]
  2 years | 48.0 [36.1 to 59.0] | 33.1 [24.1 to 42.3]
Statistical Analysis 1: Comparison: FL and MZL: Tafasitamab + Rituximab + Lenalidomide vs FL and MZL: Placebo + Rituximab + Lenalidomide; Test type: Superiority; p < 0.0001, stratified Log Rank; Hazard Ratio (HR) = 0.500, 95% CI 2-sided [0.383 to 0.653] — The hazard ratio was estimated using a stratified Cox proportional hazards model

5. Secondary Outcome: FDG-avid FL Population: Positron Emission Tomography-Complete Response (PET-CR) Rate by Investigator Assessment, Using the Lugano 2014 Criteria
Description: CR was defined as a complete metabolic response at any time after the start of treatment. Per PET, CR criteria: (1) score of 1, 2, or 3 with or without a residual mass on a 5-point scale for lymph nodes and extralymphatic sites; (2) No evidence of FDG-avid disease in bone marrow; and (3) no new lesions. PET 5-point scale: 1 = no uptake above background; 2 = uptake ≤ mediastinum; 3 = uptake > mediastinum but ≤ liver; 4 = uptake moderately > liver; 5 = uptake markedly higher than liver and/or new lesions; X = new areas of uptake unlikely to be related to lymphoma.
Time Frame: up to approximately 34 months
Population: FL FDG-avid Set: all randomized participants with FL and with a PET scan at Baseline with a resulting Deauville score of 4 or 5. Participants who did not have a post-baseline PET scan were considered to be "not assessed," but were included in the analysis. The 95% confidence intervals were calculated using the Clopper-Pearson method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 251 | 254 | 0 | 0
percentage of participants | 49.4 [43.06 to 55.76] | 39.8 [33.70 to 46.07] |  |
Statistical Analysis 1: Comparison: FL: Tafasitamab + Rituximab + Lenalidomide vs FL: Placebo + Rituximab + Lenalidomide; Test type: Superiority; p = 0.0286, stratified Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.5, 95% CI 2-sided [1.04 to 2.13] — The strata information was based on the data obtained from the interactive response technology that was used for randomization

6. Secondary Outcome: FL Population: Overall Survival
Description: Overall survival was defined as the time from randomization until death from any cause.
Time Frame: up to approximately 34 months
Population: FL Full Analysis Set. The 2-sided 95% confidence intervals were calculated using the method of Brookmeyer and Crowley with log-log transformation. Censored participants were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 273 | 275 | 0 | 0
months | NA [27.93 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants died. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants died. |  |

7. Secondary Outcome: FL Population: Kaplan-Meier Estimates of Overall Survival
Description: Overall survival was defined as the time from randomization until death from any cause. Kaplan-Meier estimates indicate the percent probability of a participant being alive at the indicated time after treatment start.
Time Frame: up to 2 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 273 | 275 | 0 | 0
percent probability
  6 months | 99.3 [97.1 to 99.8] | 96.2 [93.1 to 98.0] |  |
  12 months | 96.4 [92.8 to 98.2] | 93.7 [90.0 to 96.1] |  |
  18 months | 93.8 [89.1 to 96.5] | 90.1 [84.8 to 93.6] |  |
  2 years | 92.5 [87.0 to 95.8] | 85.5 [76.2 to 91.4] |  |
Statistical Analysis 1: Comparison: FL: Tafasitamab + Rituximab + Lenalidomide vs FL: Placebo + Rituximab + Lenalidomide; Test type: Superiority; p = 0.1061, stratified Log Rank; Hazard Ratio (HR) = 0.587, 95% CI 2-sided [0.306 to 1.128] — The hazard ratio was estimated using a stratified Cox proportional hazards model

8. Secondary Outcome: FDG-avid Overall Population: PET-CR Rate by Investigator Assessment, Using the Lugano 2014 Criteria
Description: CR was defined as a complete metabolic response at any time after the start of treatment. Per PET, CR criteria: (1) score of 1, 2, or 3 with or without a residual mass on a 5-point scale for lymph nodes and extralymphatic sites; (2) No evidence of FDG-avid disease in bone marrow; and (3) no new lesions. PET 5-point scale: 1 = no uptake above background; 2 = uptake ≤ mediastinum; 3 = uptake > mediastinum but ≤ liver; 4 = uptake moderately > liver; 5 = uptake markedly higher than liver and/or new lesions; X = new areas of uptake unlikely to be related to lymphoma. The Overall FDG-avid Set included all randomized participants with a PET scan at Baseline with a resulting Deauville score of 4 or 5.
Time Frame: up to approximately 34 months
Population: Overall FDG-avid Set. As pre-specified in the Statistical Analysis Plan, the MZL population was considered as a subpopulation of interest, not a main analysis population. The FL and MZL populations were combined for analysis into the Overall population, which was a main analysis population. Participants who did not have a post-baseline PET scan were considered to be "not assessed," but were included in the analysis. The 95% confidence intervals were calculated using the Clopper-Pearson method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FL and MZL: Tafasitamab + Rituximab + Lenalidomide | FL and MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 290 | 293
percentage of participants | 50.7 [44.78 to 56.58] | 41.3 [35.60 to 47.17]
Statistical Analysis 1: Comparison: FL and MZL: Tafasitamab + Rituximab + Lenalidomide vs FL and MZL: Placebo + Rituximab + Lenalidomide; Test type: Superiority — Only primary and key secondary endpoints were formally tested; this endpoint was not formally tested; p = 0.0221, stratified Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.5, 95% CI 2-sided [1.06 to 2.03] — [estimate comment as in outcome 5, analysis 1]

9. Secondary Outcome: FL Population: Minimal Residual Disease (MRD)-Negativity Rate (at Threshold of 10^-5) at End of Treatment
Description: The MRD-negativity rate was defined as the percentage of participants who achieved a negative MRD result in peripheral blood at the End of Treatment. The threshold used for the analysis was 10^-5 cells. MRD status was only analyzed with a threshold of ≤10^-5 cells for MRD negativity.
Time Frame: up to approximately 34 months
Population: FL MRD Blood-Evaluable Set: all participants in the Full Analysis Set with FL who received at least 1 dose of study treatment with identifiable clonality in blood samples at Cycle 1 Day 1. The 95% confidence intervals were calculated using the Clopper-Pearson method. Participants who did not have a post-baseline assessment were considered to be "not assessed," but were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 57 | 66 | 0 | 0
percentage of participants | 26.3 [15.54 to 39.66] | 18.2 [9.76 to 29.61] |  |
Statistical Analysis 1: Comparison: FL: Tafasitamab + Rituximab + Lenalidomide vs FL: Placebo + Rituximab + Lenalidomide; Test type: Superiority — Only primary and key secondary endpoints were formally tested; this endpoint was not formally tested; p = 0.4093, stratified Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.61 to 3.33] — [estimate comment as in outcome 5, analysis 1]

10. Secondary Outcome: Overall Population: MRD-negativity Rate (at Threshold of 10-5) at End of Treatment
Description: The MRD-negativity rate was defined as the percentage of participants who achieved a negative MRD result in peripheral blood at the End of Treatment. The threshold used for the analysis was 10^-5 cells. MRD status was only analyzed with a threshold of ≤10^-5 cells for MRD negativity. The Overall MRD Blood-Evaluable Set included all participants in the Full Analysis Set who received at least 1 dose of study treatment with identifiable clonality in blood samples at Cycle 1 Day 1.
Time Frame: up to approximately 34 months
Population: Overall MRD Blood-Evaluable Set. As pre-specified in the Statistical Analysis Plan, the MZL population was a subpopulation of interest, not a main analysis population. The FL and MZL populations were combined for analysis into the Overall population, which was a main analysis population. The 95% confidence intervals were calculated using the Clopper-Pearson method. Participants who did not have a post-baseline assessment were considered to be "not assessed," but were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FL and MZL: Tafasitamab + Rituximab + Lenalidomide | FL and MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 74 | 86
percentage of participants | 21.6 [12.89 to 32.72] | 15.1 [8.30 to 24.46]
Statistical Analysis 1: Comparison: FL and MZL: Tafasitamab + Rituximab + Lenalidomide vs FL and MZL: Placebo + Rituximab + Lenalidomide; Test type: Superiority — Only primary and key secondary endpoints were formally tested; this endpoint was not formally tested; p = 0.2874, stratified Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.69 to 3.47] — [estimate comment as in outcome 5, analysis 1]

11. Secondary Outcome: FL Population: Overall Response Rate (Percentage of Participants Who Achieved a CR/PR Per the Lugano Classification at Any Time During the Study But Before the First PD and Before/at the Start of a New Antilymphoma Treatment) by Investigator Assessment
Description: PET, CR: (1) score of 1 (no uptake above background), 2 (uptake ≤ mediastinum), or 3 (uptake > mediastinum but ≤ liver) with/without a residual mass for lymph nodes and extralymphatic sites (LN/ELS); (2) no evidence of FDG-avid disease in bone marrow; (3) no new lesions. PR: (1) score of 4 (uptake moderately > liver) or 5 (uptake markedly higher than liver and/or new lesions) with reduced uptake compared with Baseline and residual mass(es) of any size for LN/ELS; (2) residual uptake higher than in normal bone marrow but reduced from Baseline; (3) no new lesions. CT, CR: (1) target nodes/nodal masses regressed to ≤1.5 cm in LDi. no extra lymphatic site of disease; (2) absent nontarget lesions; (3) liver/spleen regressed to normal; (4) bone marrow normal by morphology; (5) no new lesions. PR: (1) ≥50% decrease in SPD of up to 6 target measurable nodes and extranodal sites; (2) no increase in target lesions; (3) spleen regressed by >50% in length beyond normal; (4) no new lesions.
Time Frame: up to approximately 34 months
Population: FL Full Analysis Set. The 95% confidence intervals were calculated using the Clopper-Pearson method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 273 | 275 | 0 | 0
percentage of participants | 83.5 [78.57 to 87.72] | 72.4 [66.67 to 77.56] |  |
Statistical Analysis 1: Comparison: FL: Tafasitamab + Rituximab + Lenalidomide vs FL: Placebo + Rituximab + Lenalidomide; Test type: Superiority — Only primary and key secondary endpoints were formally tested; this endpoint was not formally tested; p = 0.0014, stratified Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.0, 95% CI 2-sided [1.30 to 3.02] — [estimate comment as in outcome 5, analysis 1]

12. Secondary Outcome: Overall Population: Overall Response Rate (Percentage of Participants Who Achieved a CR/PR Per Lugano Classification at Any Time During the Study But Before the First PD and Before/at the Start of a New Antilymphoma Treatment) by Investigator Assessment
Description: as for outcome 11
Time Frame: up to approximately 34 months
Population: Overall Full Analysis Set. As pre-specified in the Statistical Analysis Plan, the MZL population was considered as a subpopulation of interest, not a main analysis population. The FL and MZL populations were combined for analysis into the Overall population, which was a main analysis population. The 95% confidence intervals were calculated using the Clopper-Pearson method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FL and MZL: Tafasitamab + Rituximab + Lenalidomide | FL and MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 326 | 328
percentage of participants | 82.8 [78.28 to 86.76] | 72.0 [66.75 to 76.75]
Statistical Analysis 1: Comparison: FL and MZL: Tafasitamab + Rituximab + Lenalidomide vs FL and MZL: Placebo + Rituximab + Lenalidomide; Test type: Superiority — Only primary and key secondary endpoints were formally tested; this endpoint was not formally tested; p = 0.0009, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.9, 95% CI 2-sided [1.29 to 2.74] — [estimate comment as in outcome 5, analysis 1]

13. Secondary Outcome: FL Population: Duration of Response (DOR; the Time From the First Tumor Response [CR or PR as Per the Lugano 2014 Classification] Until the Time of the First Documented PD or Death From Any Cause, Whichever Was Earlier) by Investigator Assessment
Description: as for outcome 11
Time Frame: up to approximately 34 months
Population: FL Full Analysis Set. The 2-sided 95% confidence intervals were calculated using the method of Brookmeyer and Crowley with log-log transformation. Only those participants who achieved an objective response (CR or PR) were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 228 | 199 | 0 | 0
months | 21.19 [19.48 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 13.60 [12.42 to 18.56] |  |

14. Secondary Outcome: FL Population: Kaplan-Meier Estimates of DOR (the Time From the First Tumor Response [CR or PR as Per the Lugano 2014 Classification] Until the Time of the First Documented PD or Death From Any Cause, Whichever Was Earlier) by Investigator Assessment
Description: as for outcome 11
Time Frame: up to 2 years
Population: FL Full Analysis Set. Only those participants who achieved an objective response (CR or PR) were analyzed. Kaplan-Meier estimates indicate the percent probability of a participant still having a CR or PR at the indicated time after treatment start. The number of participants analyzed for the Kaplan-Meier estimate at each time point refers to the total number of participants in the analysis set.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 228 | 199 | 0 | 0
percent probability
  6 months | 91.5 [86.6 to 94.6] | 77.8 [70.9 to 83.2] |  |
  12 months | 76.3 [68.4 to 82.4] | 59.1 [50.3 to 66.9] |  |
  18 months | 63.7 [53.4 to 72.2] | 42.9 [33.1 to 52.4] |  |
  2 years | 39.5 [21.4 to 57.1] | 33.3 [20.5 to 46.6] |  |
Statistical Analysis 1: Comparison: FL: Tafasitamab + Rituximab + Lenalidomide vs FL: Placebo + Rituximab + Lenalidomide; Test type: Superiority — Only primary and key secondary endpoints were formally tested; this endpoint was not formally tested; p < 0.0001, stratified Log Rank; Hazard Ratio (HR) = 0.473, 95% CI 2-sided [0.330 to 0.678] — The hazard ratio was estimated using a stratified Cox proportional hazards model

15. Secondary Outcome: Overall Population: DOR (the Time From the First Tumor Response [CR or PR as Per the Lugano 2014 Classification] Until the Time of the First Documented PD or Death From Any Cause, Whichever Was Earlier) by Investigator Assessment
Description: as for outcome 11
Time Frame: up to approximately 34 months
Population: Overall Full Analysis Set. As pre-specified in the Statistical Analysis Plan, the MZL population was considered as a subpopulation of interest, not a main analysis population. The FL and MZL populations were combined for analysis into the Overall population, which was a main analysis population. The 2-sided 95% confidence intervals were calculated using the method of Brookmeyer and Crowley with log-log transformation. Only participants who achieved an objective response (CR or PR) were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FL and MZL: Tafasitamab + Rituximab + Lenalidomide | FL and MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 270 | 236
months | 22.24 [19.81 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 17.77 [13.37 to 19.88]

16. Secondary Outcome: Overall Population: Kaplan-Meier Estimates of DOR (the Time From the First Tumor Response [CR or PR as Per the Lugano 2014 Classification] Until the Time of the First Documented PD or Death From Any Cause, Whichever Was Earlier) by Investigator Assessment
Description: as for outcome 11
Time Frame: up to 2 years
Population: Overall Full Analysis Set. Per the SAP, the MZL population was considered as a subpopulation of interest, not a main analysis population. The FL and MZL populations were combined for analysis into the Overall population (main analysis population). Participants who achieved CR or PR were analyzed. The number of participants analyzed for the Kaplan-Meier estimate at each time point refers to the total number of participants in the analysis set.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | FL and MZL: Tafasitamab + Rituximab + Lenalidomide | FL and MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 270 | 236
percent probability
  6 months | 90.8 [86.3 to 93.8] | 80.5 [74.6 to 85.3]
  12 months | 78.1 [71.4 to 83.4] | 64.4 [56.6 to 71.1]
  18 months | 66.6 [57.8 to 73.9] | 47.6 [38.4 to 56.2]
  2 years | 43.4 [27.2 to 58.6] | 35.1 [23.0 to 47.4]
Statistical Analysis 1: Comparison: FL and MZL: Tafasitamab + Rituximab + Lenalidomide vs FL and MZL: Placebo + Rituximab + Lenalidomide; Test type: Superiority — Only primary and key secondary endpoints were formally tested; this endpoint was not formally tested; p = 0.0003, stratified Log Rank; Hazard Ratio (HR) = 0.550, 95% CI 2-sided [0.397 to 0.763] — The hazard ratio was estimated using a stratified Cox proportional hazards model

17. Secondary Outcome: Overall Population: Overall Survival
Description: Overall survival was defined as the time from randomization until death from any cause.
Time Frame: up to approximately 34 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FL and MZL: Tafasitamab + Rituximab + Lenalidomide | FL and MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 326 | 328
months | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants died. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants died.

18. Secondary Outcome: Overall Population: Kaplan-Meier Estimates of Overall Survival
Description: as for outcome 7
Time Frame: up to 2 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | FL and MZL: Tafasitamab + Rituximab + Lenalidomide | FL and MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 326 | 328
percent probability
  6 months | 98.7 [96.7 to 99.5] | 96.5 [93.8 to 98.1]
  2 months | 96.4 [93.4 to 98.1] | 94.4 [91.2 to 96.5]
  18 months | 92.2 [87.7 to 95.1] | 91.7 [87.4 to 94.5]
  2 years | 90.1 [84.4 to 93.7] | 88.3 [81.1 to 92.8]
Statistical Analysis 1: Comparison: FL and MZL: Tafasitamab + Rituximab + Lenalidomide vs FL and MZL: Placebo + Rituximab + Lenalidomide; Test type: Superiority — Only primary and key secondary endpoints were formally tested; this endpoint was not formally tested; p = 0.5837, stratified Log Rank; Hazard Ratio (HR) = 0.850, 95% CI 2-sided [0.476 to 1.519] — The hazard ratio was estimated using a stratified Cox proportional hazards model

19. Secondary Outcome: FL Population: PFS by IRC Review, Using the Lugano 2014 Criteria, Defined as the Time From Randomization to the First Documented PD, or Death From Any Cause, Whichever Occurred First
Description: as for outcome 3
Time Frame: up to approximately 34 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 273 | 275 | 0 | 0
months | NA [19.29 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died. | 16.00 [13.86 to 21.06] |  |

20. Secondary Outcome: FL Population: Kaplan-Meier Estimates of PFS by IRC Review, Using the Lugano 2014 Criteria, Defined as the Time From Randomization to the First Documented PD, or Death From Any Cause, Whichever Occurred First
Description: as for outcome 2
Time Frame: up to 2 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 273 | 275 | 0 | 0
percent probability
  6 months | 94.0 [90.2 to 96.3] | 80.3 [74.9 to 84.7] |  |
  12 months | 83.1 [77.1 to 87.7] | 59.8 [52.9 to 66.1] |  |
  18 months | 67.5 [58.8 to 74.8] | 45.8 [37.3 to 53.8] |  |
  2 years | 53.9 [41.9 to 64.4] | 35.0 [24.7 to 45.6] |  |
Statistical Analysis 1: Comparison: FL: Tafasitamab + Rituximab + Lenalidomide vs FL: Placebo + Rituximab + Lenalidomide; Test type: Superiority — Only primary and key secondary endpoints were formally tested; this endpoint was not formally tested; p < 0.0001, stratified Log Rank; Hazard Ratio (HR) = 0.407, 95% CI 2-sided [0.294 to 0.563] — The hazard ratio was estimated using a stratified Cox proportional hazards model

21. Secondary Outcome: Overall Population: PFS by IRC Review, Using the Lugano 2014 Criteria, Defined as the Time From Randomization to the First Documented PD, or Death From Any Cause, Whichever Occurred First
Description: as for outcome 3
Time Frame: up to approximately 34 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FL and MZL: Tafasitamab + Rituximab + Lenalidomide | FL and MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 326 | 328
months | NA [22.08 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died. | 20.73 [15.38 to 23.10]

22. Secondary Outcome: Overall Population: Kaplan-Meier Estimates of PFS by IRC Review, Using the Lugano 2014 Criteria, Defined as the Time From Randomization to the First Documented PD, or Death From Any Cause, Whichever Occurred First
Description: as for outcome 2
Time Frame: up to 2 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | FL and MZL: Tafasitamab + Rituximab + Lenalidomide | FL and MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 326 | 328
percent probability
  6 months | 93.9 [90.4 to 96.1] | 82.5 [77.7 to 86.4]
  12 months | 84.5 [79.2 to 88.5] | 63.7 [57.5 to 69.3]
  18 months | 68.9 [61.1 to 75.4] | 52.0 [44.5 to 59.0]
  2 years | 56.0 [45.1 to 65.6] | 38.8 [28.3 to 49.1]
Statistical Analysis 1: Comparison: FL and MZL: Tafasitamab + Rituximab + Lenalidomide vs FL and MZL: Placebo + Rituximab + Lenalidomide; Test type: Superiority — Only primary and key secondary endpoints were formally tested; this endpoint was not formally tested; p < 0.0001, stratified Log Rank; Hazard Ratio (HR) = 0.481, 95% CI 2-sided [0.357 to 0.647] — The hazard ratio was estimated using a stratified Cox proportional hazards model

23. Secondary Outcome: FL Population: Overall Response Rate (Percentage of Participants Who Achieved a CR/PR Per the Lugano Classification at Any Time During the Study But Before the First PD and Before/at the Start of a New Antilymphoma Treatment) by IRC Review
Description: as for outcome 11
Time Frame: up to approximately 34 months
Population: FL Full Analysis Set. The 95% confidence intervals were calculated using the Clopper-Pearson method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 273 | 275 | 0 | 0
percentage of participants | 85.7 [80.99 to 89.64] | 73.5 [67.82 to 78.58] |  |
Statistical Analysis 1: Comparison: FL: Tafasitamab + Rituximab + Lenalidomide vs FL: Placebo + Rituximab + Lenalidomide; Test type: Superiority — Only primary and key secondary endpoints were formally tested; this endpoint was not formally tested; p = 0.0003, stratified Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.2, 95% CI 2-sided [1.43 to 3.43] — [estimate comment as in outcome 5, analysis 1]

24. Secondary Outcome: Overall Population: Overall Response Rate (Percentage of Participants Who Achieved a CR/PR Per Lugano Classification at Any Time During the Study But Before the First PD and Before/at the Start of a New Antilymphoma Treatment) by IRC Review
Description: as for outcome 11
Time Frame: up to approximately 34 months
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FL and MZL: Tafasitamab + Rituximab + Lenalidomide | FL and MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 326 | 328
percentage of participants | 83.7 [79.28 to 87.58] | 72.6 [67.39 to 77.32]
Statistical Analysis 1: Comparison: FL and MZL: Tafasitamab + Rituximab + Lenalidomide vs FL and MZL: Placebo + Rituximab + Lenalidomide; Test type: Superiority — Only primary and key secondary endpoints were formally tested; this endpoint was not formally tested; p = 0.0005, stratified Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.0, 95% CI 2-sided [1.33 to 2.86] — [estimate comment as in outcome 5, analysis 1]

25. Secondary Outcome: FL Population: DOR the Time From the First Tumor Response [CR or PR as Per the Lugano 2014 Classification] Until the Time of the First Documented PD or Death From Any Cause, Whichever Was Earlier) by IRC Review
Description: as for outcome 11
Time Frame: up to approximately 34 months
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 234 | 202 | 0 | 0
months | NA [19.02 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died. | 18.23 [12.94 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. |  |

26. Secondary Outcome: FL Population: Kaplan-Meier Estimates of DOR (the Time From the First Tumor Response [CR or PR as Per the Lugano 2014 Classification] Until the Time of the First Documented PD or Death From Any Cause, Whichever Was Earlier) by IRC Review
Description: as for outcome 11
Time Frame: up to 2 years
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 234 | 202 | 0 | 0
percent probability
  6 months | 92.4 [87.6 to 95.3] | 78.7 [71.8 to 84.0] |  |
  12 months | 78.8 [70.9 to 84.8] | 61.4 [52.4 to 69.3] |  |
  18 months | 64.3 [53.1 to 73.5] | 52.2 [41.7 to 61.7] |  |
  2 years | 58.2 [44.9 to 69.4] | 35.5 [21.3 to 50.0] |  |
Statistical Analysis 1: Comparison: FL: Tafasitamab + Rituximab + Lenalidomide vs FL: Placebo + Rituximab + Lenalidomide; Test type: Superiority — Only primary and key secondary endpoints were formally tested; this endpoint was not formally tested; p < 0.0001, stratified Log Rank; Hazard Ratio (HR) = 0.461, 95% CI 2-sided [0.312 to 0.681] — The hazard ratio was estimated using a stratified Cox proportional hazards model

27. Secondary Outcome: Overall Population: DOR (the Time From the First Tumor Response [CR or PR as Per the Lugano 2014 Classification] Until the Time of the First Documented PD or Death From Any Cause, Whichever Was Earlier) by IRC Review
Description: as for outcome 11
Time Frame: up to approximately 34 months
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FL and MZL: Tafasitamab + Rituximab + Lenalidomide | FL and MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 273 | 238
months | NA [19.52 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died. | 18.83 [16.89 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died.

28. Secondary Outcome: Overall Population: Kaplan-Meier Estimates of DOR (the Time From the First Tumor Response [CR or PR as Per the Lugano 2014 Classification] Until the Time of the First Documented PD or Death From Any Cause, Whichever Was Earlier) by IRC Review
Description: as for outcome 11
Time Frame: up to 2 years
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | FL and MZL: Tafasitamab + Rituximab + Lenalidomide | FL and MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 273 | 238
percent probability
  6 months | 93.1 [88.9 to 95.7] | 81.5 [75.5 to 86.2]
  12 months | 80.0 [73.0 to 85.3] | 65.6 [57.6 to 72.5]
  18 months | 65.7 [55.8 to 73.8] | 56.5 [46.9 to 65.0]
  2 years | 56.0 [41.5 to 68.2] | 40.9 [27.8 to 53.6]
Statistical Analysis 1: Comparison: FL and MZL: Tafasitamab + Rituximab + Lenalidomide vs FL and MZL: Placebo + Rituximab + Lenalidomide; Test type: Superiority — Only primary and key secondary endpoints were formally tested; this endpoint was not formally tested; p = 0.7469, stratified Log Rank; Hazard Ratio (HR) = 1.192, 95% CI 2-sided [0.409 to 3.475] — The hazard ratio was estimated using a stratified Cox proportional hazards model

29. Secondary Outcome: FL Population: EORTC QLQ-C30 Scores at Baseline and End of Treatment
Description: The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-30 (EORTC QLQ-C30) version 3 is a 30-item scale composed of both multi-item scales and single-item measures. These include 5 functional scales (physical functioning, role, cognitive functioning, emotional functioning, and social functioning), 3 symptom scales (fatigue, pain, and nausea/vomiting), a global health status scale, and 6 single items (constipation, diarrhea, sleep, dyspnea, appetite, financial). All scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Therefore, a high score for a functional scale represents a high/healthy level of functioning and a high score for the global health status/QoL represents a high QoL. A high score for a symptom scale/item represents a high level of symptomatology/problems. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: up to approximately 34 months
Population: FL Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 273 | 275 | 0 | 0
scores on a scale
  Baseline, Global Health Status: number analyzed (Participants) | 266 | 266 | 0 | 0
  Baseline, Global Health Status | 68.6 (20.44) | 68.6 (21.93) |  |
  End of Treatment, Global Health Status: number analyzed (Participants) | 186 | 186 | 0 | 0
  End of Treatment, Global Health Status | 67.7 (21.37) | 67.5 (21.00) |  |
  Baseline, Physical Functioning: number analyzed (Participants) | 266 | 267 | 0 | 0
  Baseline, Physical Functioning | 84.7 (17.44) | 84.1 (19.54) |  |
  End of Treatment, Physical Functioning: number analyzed (Participants) | 186 | 186 | 0 | 0
  End of Treatment, Physical Functioning | 80.1 (21.02) | 81.0 (22.67) |  |
  Baseline, Role Functioning: number analyzed (Participants) | 266 | 267 | 0 | 0
  Baseline, Role Functioning | 83.1 (22.72) | 82.8 (24.72) |  |
  End of Treatment, Role Functioning: number analyzed (Participants) | 186 | 186 | 0 | 0
  End of Treatment, Role Functioning | 77.3 (26.75) | 76.2 (29.09) |  |
  Baseline, Emotional Functioning: number analyzed (Participants) | 265 | 267 | 0 | 0
  Baseline, Emotional Functioning | 79.2 (19.04) | 79.2 (19.03) |  |
  End of Treatment, Emotional Functioning: number analyzed (Participants) | 186 | 186 | 0 | 0
  End of Treatment, Emotional Functioning | 79.0 (20.79) | 79.1 (21.36) |  |
  Baseline, Cognitive Functioning: number analyzed (Participants) | 266 | 266 | 0 | 0
  Baseline, Cognitive Functioning | 88.0 (19.06) | 87.0 (17.25) |  |
  End of Treatment, Cognitive Functioning: number analyzed (Participants) | 186 | 186 | 0 | 0
  End of Treatment, Cognitive Functioning | 83.6 (20.45) | 82.4 (21.03) |  |
  Baseline, Social Functioning: number analyzed (Participants) | 266 | 267 | 0 | 0
  Baseline, Social Functioning | 84.7 (19.77) | 83.4 (22.50) |  |
  End of Treatment, Social Functioning: number analyzed (Participants) | 186 | 186 | 0 | 0
  End of Treatment, Social Functioning | 79.8 (25.77) | 81.2 (23.63) |  |
  Baseline, Fatigue: number analyzed (Participants) | 266 | 267 | 0 | 0
  Baseline, Fatigue | 27.0 (23.43) | 26.9 (24.71) |  |
  End of Treatment, Fatigue: number analyzed (Participants) | 186 | 186 | 0 | 0
  End of Treatment, Fatigue | 30.5 (25.06) | 31.0 (25.39) |  |
  Baseline, Nausea and Vomiting: number analyzed (Participants) | 266 | 267 | 0 | 0
  Baseline, Nausea and Vomiting | 2.7 (7.91) | 2.9 (9.62) |  |
  End of Treatment, Nausea and Vomiting: number analyzed (Participants) | 186 | 186 | 0 | 0
  End of Treatment, Nausea and Vomiting | 3.2 (10.61) | 3.7 (11.61) |  |
  Baseline, Pain: number analyzed (Participants) | 266 | 267 | 0 | 0
  Baseline, Pain | 16.0 (21.06) | 17.6 (23.97) |  |
  End of Treatment, Pain: number analyzed (Participants) | 186 | 186 | 0 | 0
  End of Treatment, Pain | 17.8 (23.40) | 20.2 (27.15) |  |
  Baseline, Dyspnea: number analyzed (Participants) | 266 | 267 | 0 | 0
  Baseline, Dyspnea | 14.3 (23.79) | 16.0 (24.88) |  |
  End of Treatment, Dyspnea: number analyzed (Participants) | 186 | 186 | 0 | 0
  End of Treatment, Dyspnea | 15.7 (23.54) | 17.5 (25.01) |  |
  Baseline, Sleep: number analyzed (Participants) | 266 | 267 | 0 | 0
  Baseline, Sleep | 26.1 (27.86) | 25.3 (27.50) |  |
  End of Treatment, Sleep: number analyzed (Participants) | 186 | 186 | 0 | 0
  End of Treatment, Sleep | 25.0 (28.67) | 27.7 (27.75) |  |
  Baseline, Appetite Loss: number analyzed (Participants) | 266 | 267 | 0 | 0
  Baseline, Appetite Loss | 10.2 (23.21) | 11.4 (20.45) |  |
  End of Treatment, Appetite Loss: number analyzed (Participants) | 186 | 186 | 0 | 0
  End of Treatment, Appetite Loss | 12.5 (23.46) | 12.3 (22.60) |  |
  Baseline, Constipation: number analyzed (Participants) | 266 | 267 | 0 | 0
  Baseline, Constipation | 9.2 (19.55) | 11.4 (20.86) |  |
  End of Treatment, Constipation: number analyzed (Participants) | 186 | 186 | 0 | 0
  End of Treatment, Constipation | 11.4 (22.16) | 12.5 (24.96) |  |
  Baseline, Diarrhea: number analyzed (Participants) | 266 | 267 | 0 | 0
  Baseline, Diarrhea | 7.0 (14.98) | 5.7 (15.00) |  |
  End of Treatment, Diarrhea: number analyzed (Participants) | 186 | 186 | 0 | 0
  End of Treatment, Diarrhea | 12.7 (24.74) | 12.5 (21.86) |  |
  Baseline, Financial Difficulties: number analyzed (Participants) | 266 | 267 | 0 | 0
  Baseline, Financial Difficulties | 12.2 (23.34) | 12.0 (20.37) |  |
  End of Treatment, Financial Difficulties: number analyzed (Participants) | 186 | 186 | 0 | 0
  End of Treatment, Financial Difficulties | 11.8 (21.70) | 12.7 (22.69) |  |

30. Secondary Outcome: Overall Population: EORTC QLQ-C30 Scores at Baseline and End of Treatment
Description: as for outcome 29
Time Frame: up to approximately 34 months
Population: Overall Full Analysis Set. As pre-specified in the Statistical Analysis Plan, the MZL population was considered as a subpopulation of interest, not a main analysis population. The FL and MZL populations were combined for analysis into the Overall population, which was a main analysis population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | FL and MZL: Tafasitamab + Rituximab + Lenalidomide | FL and MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 326 | 328
scores on a scale
  Baseline, Global Health Status: number analyzed (Participants) | 317 | 317
  Baseline, Global Health Status | 68.5 (20.59) | 67.3 (22.67)
  End of Treatment, Global Health Status: number analyzed (Participants) | 229 | 228
  End of Treatment, Global Health Status | 68.2 (20.96) | 66.6 (21.24)
  Baseline, Physical Functioning: number analyzed (Participants) | 317 | 318
  Baseline, Physical Functioning | 83.2 (18.07) | 82.8 (20.20)
  End of Treatment, Physical Functioning: number analyzed (Participants) | 229 | 228
  End of Treatment, Physical Functioning | 80.3 (21.21) | 80.2 (22.34)
  Baseline, Role Functioning: number analyzed (Participants) | 317 | 318
  Baseline, Role Functioning | 82.2 (23.85) | 81.1 (25.48)
  End of Treatment, Role Functioning: number analyzed (Participants) | 229 | 228
  End of Treatment, Role Functioning | 78.1 (26.41) | 75.5 (28.94)
  Baseline, Emotional Functioning: number analyzed (Participants) | 316 | 318
  Baseline, Emotional Functioning | 79.5 (19.36) | 78.8 (19.31)
  End of Treatment, Emotional Functioning: number analyzed (Participants) | 229 | 228
  End of Treatment, Emotional Functioning | 80.2 (20.55) | 79.1 (21.22)
  Baseline, Cognitive Functioning: number analyzed (Participants) | 317 | 317
  Baseline, Cognitive Functioning | 87.6 (18.79) | 86.8 (17.03)
  End of Treatment, Cognitive Functioning: number analyzed (Participants) | 229 | 228
  End of Treatment, Cognitive Functioning | 83.6 (20.09) | 82.6 (20.87)
  Baseline, Social functioning: number analyzed (Participants) | 317 | 318
  Baseline, Social functioning | 84.6 (19.94) | 82.3 (23.47)
  End of Treatment, Social Functioning: number analyzed (Participants) | 229 | 228
  End of Treatment, Social Functioning | 81.0 (25.37) | 81.5 (22.86)
  Baseline, Fatigue: number analyzed (Participants) | 317 | 318
  Baseline, Fatigue | 28.5 (24.55) | 28.3 (25.77)
  End of Treatment, Fatigue: number analyzed (Participants) | 229 | 228
  End of Treatment, Fatigue | 30.1 (24.52) | 31.0 (25.08)
  Baseline, Nausea and Vomiting: number analyzed (Participants) | 317 | 318
  Baseline, Nausea and Vomiting | 2.8 (9.31) | 2.9 (9.16)
  End of Treatment, Nausea and Vomiting: number analyzed (Participants) | 229 | 228
  End of Treatment, Nausea and Vomiting | 3.4 (10.56) | 4.1 (12.34)
  Baseline, Pain: number analyzed (Participants) | 317 | 318
  Baseline, Pain | 17.2 (22.35) | 17.8 (23.89)
  End of Treatment, Pain: number analyzed (Participants) | 229 | 228
  End of Treatment, Pain | 17.9 (23.73) | 19.7 (26.42)
  Baseline, Dyspnea: number analyzed (Participants) | 317 | 318
  Baseline, Dyspnea | 15.8 (24.79) | 17.2 (26.27)
  End of Treatment, Dyspnea: number analyzed (Participants) | 229 | 228
  End of Treatment, Dyspnea | 16.2 (24.50) | 18.5 (25.80)
  Baseline, Sleep: number analyzed (Participants) | 317 | 318
  Baseline, Sleep | 27.8 (29.41) | 25.9 (27.20)
  End of Treatment, Sleep: number analyzed (Participants) | 229 | 228
  End of Treatment, Sleep | 25.7 (29.33) | 26.8 (27.81)
  Baseline, Appetite Loss: number analyzed (Participants) | 317 | 318
  Baseline, Appetite Loss | 11.2 (24.51) | 11.5 (20.31)
  End of Treatment, Appetite Loss: number analyzed (Participants) | 229 | 229
  End of Treatment, Appetite Loss | 12.6 (23.35) | 12.9 (23.40)
  Baseline, Constipation: number analyzed (Participants) | 317 | 318
  Baseline, Constipation | 9.8 (20.70) | 10.8 (20.46)
  End of Treatment, Constipation: number analyzed (Participants) | 229 | 228
  End of Treatment, Constipation | 11.7 (23.37) | 12.7 (24.62)
  Baseline, Diarrhea: number analyzed (Participants) | 317 | 318
  Baseline, Diarrhea | 7.5 (16.02) | 5.6 (14.81)
  End of Treatment, Diarrhea: number analyzed (Participants) | 229 | 228
  End of Treatment, Diarrhea | 12.5 (23.95) | 13.7 (23.53)
  Baseline, Financial Difficulties: number analyzed (Participants) | 317 | 318
  Baseline, Financial Difficulties | 11.9 (22.58) | 12.5 (21.20)
  End of Treatment, Financial Difficulties: number analyzed (Participants) | 229 | 228
  End of Treatment, Financial Difficulties | 11.4 (21.12) | 12.2 (21.99)

31. Secondary Outcome: FL Population: Health State EQ-5D-5L Scores at Baseline and End of Treatment
Description: The EQ-5D-5L contains a participant-reported score regarding health state measured on a visual analog scale (scores range from 0 [worst imaginable health state] to 100 [best imaginable health state]), and 5 questions on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The 5 questions have 5 response levels: 1, no problems; 2, slight problems; 3, moderate problems; 4, severe problems; and 5, unable to/extreme problems.
Time Frame: up to approximately 34 months
Population: FL Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 264 | 264 | 0 | 0
scores on a scale
  Baseline | 72.5 (18.15) | 73.6 (19.13) |  |
  End of Treatment: number analyzed (Participants) | 186 | 186 | 0 | 0
  End of Treatment | 73.7 (18.21) | 72.5 (19.17) |  |

32. Secondary Outcome: Overall Population: Health State EQ-5D-5L Scores at Baseline and End of Treatment
Description: as for outcome 31
Time Frame: up to approximately 34 months
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | FL and MZL: Tafasitamab + Rituximab + Lenalidomide | FL and MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 315 | 313
scores on a scale
  Baseline | 72.2 (18.78) | 72.6 (19.67)
  End of Treatment: number analyzed (Participants) | 228 | 228
  End of Treatment | 74.2 (18.37) | 72.0 (19.21)

33. Secondary Outcome: FL Population: Number of Participants With the Indicated Scores for the Five EQ-5D-5L Domains/Questions at Baseline and End of Treatment
Description: as for outcome 31
Time Frame: up to approximately 34 months
Population: FL Full Analysis Set. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 273 | 275 | 0 | 0
Participants
  Baseline, Mobility, Score 1: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Mobility, Score 1 | 185 | 198 |  |
  Baseline, Mobility, Score 2: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Mobility, Score 2 | 58 | 34 |  |
  Baseline, Mobility, Score 3: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Mobility, Score 3 | 16 | 25 |  |
  Baseline, Mobility, Score 4: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Mobility, Score 4 | 4 | 8 |  |
  Baseline, Mobility, Score 5: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Mobility, Score 5 | 1 | 0 |  |
  End of Treatment, Mobility, Score 1: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Mobility, Score 1 | 122 | 126 |  |
  End of Treatment, Mobility, Score 2: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Mobility, Score 2 | 39 | 34 |  |
  End of Treatment, Mobility, Score 3: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Mobility, Score 3 | 14 | 17 |  |
  End of Treatment, Mobility, Score 4: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Mobility, Score 4 | 9 | 9 |  |
  End of Treatment, Mobility, Score 5: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Mobility, Score 5 | 2 | 1 |  |
  Baseline, Self-care, Score 1: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Self-care, Score 1 | 250 | 243 |  |
  Baseline, Self-care, Score 2: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Self-care, Score 2 | 9 | 16 |  |
  Baseline, Self-care, Score 3: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Self-care, Score 3 | 3 | 4 |  |
  Baseline, Self-care, Score 4: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Self-care, Score 4 | 1 | 1 |  |
  Baseline, Self-care, Score 5: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Self-care, Score 5 | 1 | 1 |  |
  End of Treatment, Self-care, Score 1: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Self-care, Score 1 | 165 | 166 |  |
  End of Treatment, Self-care, Score 2: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Self-care, Score 2 | 12 | 9 |  |
  End of Treatment, Self-care, Score 3: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Self-care, Score 3 | 6 | 7 |  |
  End of Treatment, Self-care, Score 4: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Self-care, Score 4 | 3 | 5 |  |
  End of Treatment, Self-care, Score 5: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Self-care, Score 5 | 0 | 0 |  |
  Baseline, Usual Activities, Score 1: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Usual Activities, Score 1 | 179 | 184 |  |
  Baseline, Usual Activities, Score 2: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Usual Activities, Score 2 | 59 | 50 |  |
  Baseline, Usual Activities, Score 3: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Usual Activities, Score 3 | 17 | 26 |  |
  Baseline, Usual Activities, Score 4: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Usual Activities, Score 4 | 4 | 4 |  |
  Baseline, Usual Activities, Score 5: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Usual Activities, Score 5 | 5 | 1 |  |
  End of Treatment, Usual Activities, Score 1: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Usual Activities, Score 1 | 107 | 114 |  |
  End of Treatment, Usual Activities, Score 2: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Usual Activities, Score 2 | 58 | 47 |  |
  End of Treatment, Usual Activities, Score 3: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Usual Activities, Score 3 | 13 | 16 |  |
  End of Treatment, Usual Activities, Score 4: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Usual Activities, Score 4 | 7 | 5 |  |
  End of Treatment, Usual Activities, Score 5: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Usual Activities, Score 5 | 1 | 5 |  |
  Baseline, Pain/Discomfort, Score 1: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Pain/Discomfort, Score 1 | 144 | 141 |  |
  Baseline, Pain/Discomfort, Score 2: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Pain/Discomfort, Score 2 | 92 | 82 |  |
  Baseline, Pain/Discomfort, Score 3: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Pain/Discomfort, Score 3 | 25 | 34 |  |
  Baseline, Pain/Discomfort, Score 4: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Pain/Discomfort, Score 4 | 2 | 7 |  |
  Baseline, Pain/Discomfort, Score 5: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Pain/Discomfort, Score 5 | 1 | 1 |  |
  End of Treatment, Pain/Discomfort, Score 1: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Pain/Discomfort, Score 1 | 106 | 104 |  |
  End of Treatment, Pain/Discomfort, Score 2: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Pain/Discomfort, Score 2 | 55 | 51 |  |
  End of Treatment, Pain/Discomfort, Score 3: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Pain/Discomfort, Score 3 | 17 | 21 |  |
  End of Treatment, Pain/Discomfort, Score 4: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Pain/Discomfort, Score 4 | 8 | 8 |  |
  End of Treatment, Pain/Discomfort, Score 5: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Pain/Discomfort, Score 5 | 0 | 3 |  |
  Baseline, Anxiety/Depression, Score 1: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Anxiety/Depression, Score 1 | 138 | 152 |  |
  Baseline, Anxiety/Depression, Score 2: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Anxiety/Depression, Score 2 | 98 | 79 |  |
  Baseline, Anxiety/Depression, Score 3: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Anxiety/Depression, Score 3 | 22 | 26 |  |
  Baseline, Anxiety/Depression, Score 4: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Anxiety/Depression, Score 4 | 5 | 7 |  |
  Baseline, Anxiety/Depression, Score 5: number analyzed (Participants) | 264 | 265 | 0 | 0
  Baseline, Anxiety/Depression, Score 5 | 1 | 1 |  |
  End of Treatment, Anxiety/Depression, Score 1: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Anxiety/Depression, Score 1 | 107 | 103 |  |
  End of Treatment, Anxiety/Depression, Score 2: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Anxiety/Depression, Score 2 | 58 | 60 |  |
  End of Treatment, Anxiety/Depression, Score 3: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Anxiety/Depression, Score 3 | 18 | 20 |  |
  End of Treatment, Anxiety/Depression, Score 4: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Anxiety/Depression, Score 4 | 1 | 4 |  |
  End of Treatment, Anxiety/Depression, Score 5: number analyzed (Participants) | 186 | 187 | 0 | 0
  End of Treatment, Anxiety/Depression, Score 5 | 2 | 0 |  |

34. Secondary Outcome: Overall Population: Number of Participants With the Indicated Scores for the Five EQ-5D-5L Domains/Questions at Baseline and End of Treatment
Description: as for outcome 31
Time Frame: up to approximately 34 months
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | FL and MZL: Tafasitamab + Rituximab + Lenalidomide | FL and MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 326 | 328
Participants
  Baseline, Mobility, Score 1: number analyzed (Participants) | 315 | 314
  Baseline, Mobility, Score 1 | 212 | 226
  Baseline, Mobility, Score 2: number analyzed (Participants) | 315 | 314
  Baseline, Mobility, Score 2 | 68 | 47
  Baseline, Mobility, Score 3: number analyzed (Participants) | 315 | 314
  Baseline, Mobility, Score 3 | 24 | 30
  Baseline, Mobility, Score 4: number analyzed (Participants) | 315 | 314
  Baseline, Mobility, Score 4 | 10 | 11
  Baseline, Mobility, Score 5: number analyzed (Participants) | 315 | 314
  Baseline, Mobility, Score 5 | 1 | 0
  End of Treatment, Mobility, Score 1: number analyzed (Participants) | 228 | 229
  End of Treatment, Mobility, Score 1 | 149 | 149
  End of Treatment, Mobility, Score 2: number analyzed (Participants) | 228 | 229
  End of Treatment, Mobility, Score 2 | 46 | 47
  End of Treatment, Mobility, Score 3: number analyzed (Participants) | 228 | 229
  End of Treatment, Mobility, Score 3 | 17 | 22
  End of Treatment, Mobility, Score 4: number analyzed (Participants) | 228 | 229
  End of Treatment, Mobility, Score 4 | 13 | 10
  End of Treatment, Mobility, Score 5: number analyzed (Participants) | 228 | 229
  End of Treatment, Mobility, Score 5 | 3 | 1
  Baseline, Self-care, Score 1: number analyzed (Participants) | 315 | 314
  Baseline, Self-care, Score 1 | 294 | 284
  Baseline, Self-care, Score 2: number analyzed (Participants) | 315 | 314
  Baseline, Self-care, Score 2 | 12 | 22
  Baseline, Self-care, Score 3: number analyzed (Participants) | 315 | 314
  Baseline, Self-care, Score 3 | 4 | 6
  Baseline, Self-care, Score 4: number analyzed (Participants) | 315 | 314
  Baseline, Self-care, Score 4 | 2 | 1
  Baseline, Self-care, Score 5: number analyzed (Participants) | 315 | 314
  Baseline, Self-care, Score 5 | 3 | 1
  End of Treatment, Self-care, Score 1: number analyzed (Participants) | 228 | 229
  End of Treatment, Self-care, Score 1 | 198 | 202
  End of Treatment, Self-care, Score 2: number analyzed (Participants) | 228 | 229
  End of Treatment, Self-care, Score 2 | 15 | 15
  End of Treatment, Self-care, Score 3: number analyzed (Participants) | 228 | 229
  End of Treatment, Self-care, Score 3 | 9 | 7
  End of Treatment, Self-care, Score 4: number analyzed (Participants) | 228 | 229
  End of Treatment, Self-care, Score 4 | 5 | 5
  End of Treatment, Self-care, Score 5: number analyzed (Participants) | 228 | 229
  End of Treatment, Self-care, Score 5 | 1 | 0
  Baseline, Usual Activities, Score 1: number analyzed (Participants) | 315 | 314
  Baseline, Usual Activities, Score 1 | 207 | 208
  Baseline, Usual Activities, Score 2: number analyzed (Participants) | 315 | 314
  Baseline, Usual Activities, Score 2 | 74 | 64
  Baseline, Usual Activities, Score 3: number analyzed (Participants) | 315 | 314
  Baseline, Usual Activities, Score 3 | 23 | 33
  Baseline, Usual Activities, Score 4: number analyzed (Participants) | 315 | 314
  Baseline, Usual Activities, Score 4 | 6 | 5
  Baseline, Usual Activities, Score 5: number analyzed (Participants) | 315 | 314
  Baseline, Usual Activities, Score 5 | 5 | 4
  End of Treatment, Usual Activities, Score 1: number analyzed (Participants) | 228 | 229
  End of Treatment, Usual Activities, Score 1 | 133 | 135
  End of Treatment, Usual Activities, Score 2: number analyzed (Participants) | 228 | 229
  End of Treatment, Usual Activities, Score 2 | 68 | 62
  End of Treatment, Usual Activities, Score 3: number analyzed (Participants) | 228 | 229
  End of Treatment, Usual Activities, Score 3 | 15 | 21
  End of Treatment, Usual Activities, Score 4: number analyzed (Participants) | 228 | 229
  End of Treatment, Usual Activities, Score 4 | 11 | 6
  End of Treatment, Usual Activities, Score 5: number analyzed (Participants) | 228 | 229
  End of Treatment, Usual Activities, Score 5 | 1 | 5
  Baseline, Pain/Discomfort, Score 1: number analyzed (Participants) | 315 | 314
  Baseline, Pain/Discomfort, Score 1 | 168 | 161
  Baseline, Pain/Discomfort, Score 2: number analyzed (Participants) | 315 | 314
  Baseline, Pain/Discomfort, Score 2 | 108 | 104
  Baseline, Pain/Discomfort, Score 3: number analyzed (Participants) | 315 | 314
  Baseline, Pain/Discomfort, Score 3 | 35 | 40
  Baseline, Pain/Discomfort, Score 4: number analyzed (Participants) | 315 | 314
  Baseline, Pain/Discomfort, Score 4 | 3 | 8
  Baseline, Pain/Discomfort, Score 5: number analyzed (Participants) | 315 | 314
  Baseline, Pain/Discomfort, Score 5 | 1 | 1
  End of Treatment, Pain/Discomfort, Score 1: number analyzed (Participants) | 228 | 229
  End of Treatment, Pain/Discomfort, Score 1 | 129 | 124
  End of Treatment, Pain/Discomfort, Score 2: number analyzed (Participants) | 228 | 229
  End of Treatment, Pain/Discomfort, Score 2 | 68 | 70
  End of Treatment, Pain/Discomfort, Score 3: number analyzed (Participants) | 228 | 229
  End of Treatment, Pain/Discomfort, Score 3 | 21 | 23
  End of Treatment, Pain/Discomfort, Score 4: number analyzed (Participants) | 228 | 229
  End of Treatment, Pain/Discomfort, Score 4 | 10 | 9
  End of Treatment, Pain/Discomfort, Score 5: number analyzed (Participants) | 228 | 229
  End of Treatment, Pain/Discomfort, Score 5 | 0 | 3
  Baseline, Anxiety/Depression, Score 1: number analyzed (Participants) | 315 | 314
  Baseline, Anxiety/Depression, Score 1 | 173 | 177
  Baseline, Anxiety/Depression, Score 2: number analyzed (Participants) | 315 | 314
  Baseline, Anxiety/Depression, Score 2 | 110 | 98
  Baseline, Anxiety/Depression, Score 3: number analyzed (Participants) | 315 | 314
  Baseline, Anxiety/Depression, Score 3 | 25 | 30
  Baseline, Anxiety/Depression, Score 4: number analyzed (Participants) | 315 | 314
  Baseline, Anxiety/Depression, Score 4 | 6 | 8
  Baseline, Anxiety/Depression, Score 5: number analyzed (Participants) | 315 | 314
  Baseline, Anxiety/Depression, Score 5 | 1 | 1
  End of Treatment, Anxiety/Depression, Score 1: number analyzed (Participants) | 228 | 229
  End of Treatment, Anxiety/Depression, Score 1 | 136 | 126
  End of Treatment, Anxiety/Depression, Score 2: number analyzed (Participants) | 228 | 229
  End of Treatment, Anxiety/Depression, Score 2 | 68 | 74
  End of Treatment, Anxiety/Depression, Score 3: number analyzed (Participants) | 228 | 229
  End of Treatment, Anxiety/Depression, Score 3 | 20 | 24
  End of Treatment, Anxiety/Depression, Score 4: number analyzed (Participants) | 228 | 229
  End of Treatment, Anxiety/Depression, Score 4 | 2 | 5
  End of Treatment, Anxiety/Depression, Score 5: number analyzed (Participants) | 228 | 229
  End of Treatment, Anxiety/Depression, Score 5 | 2 | 0

35. Secondary Outcome: FL Population: Functional Assessment of Cancer Treatment-Lymphoma (FACT-Lym) Scores at Baseline and End of Treatment
Description: The FACT-Lymphoma (v4) is composed of 42 items with a 5-point Likert-type scale and 5 subscales. Physical well-being (PWB) subscale: 7 items measured on 0- to 4-point scale; total score = 0-28. Social/family well-being (SWB) subscale: 7 items measured on 0- to 4-point scale; total score = 0-28. Emotional well-being (EWB) subscale: 6 items measured on 0- to 4-point scale; total score = 0-24. Functional well-being (FWB) subscale: 7 items measured on 0- to 4-point scale; total score = 0-28. Lymphoma (LymS) subscale includes 15 items; total score = 0-60. Three total scores can be derived by adding the subscales: FACT-Lymphoma Trial Outcome Index (TOI): (PWB score) + (FWB score) + (LymS score); total score = 0-116. FACT-G total score: (PWB score) + (SWB score) + (EWB score) + (FWB score); total score = 0-108. FACT-Lymphoma total score: (PWB score) + (SWB score) + (EWB score) + (FWB score) + (LymS score); total score = 0-168. The higher the score, the better the quality of life.
Time Frame: up to approximately 34 months
Population: FL Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | FL: Tafasitamab + Rituximab + Lenalidomide | FL: Placebo + Rituximab + Lenalidomide | MZL: Tafasitamab + Rituximab + Lenalidomide | MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 273 | 275 | 0 | 0
scores on a scale
  Baseline, PWB subscale: number analyzed (Participants) | 259 | 263 | 0 | 0
  Baseline, PWB subscale | 24.0 (4.26) | 24.3 (4.07) |  |
  End of Treatment, PWB subscale: number analyzed (Participants) | 184 | 183 | 0 | 0
  End of Treatment, PWB subscale | 23.5 (4.68) | 23.2 (5.42) |  |
  Baseline, SWB subscale: number analyzed (Participants) | 260 | 264 | 0 | 0
  Baseline, SWB subscale | 20.9 (5.82) | 20.5 (5.92) |  |
  End of Treatment, SWB subscale: number analyzed (Participants) | 182 | 181 | 0 | 0
  End of Treatment, SWB subscale | 19.9 (5.95) | 19.9 (5.31) |  |
  Baseline, EWB subscale: number analyzed (Participants) | 261 | 265 | 0 | 0
  Baseline, EWB subscale | 18.2 (4.21) | 18.3 (4.06) |  |
  End of Treatment, EWB subscale: number analyzed (Participants) | 184 | 183 | 0 | 0
  End of Treatment, EWB subscale | 18.3 (4.39) | 18.1 (4.80) |  |
  Baseline, FWB subscale: number analyzed (Participants) | 261 | 265 | 0 | 0
  Baseline, FWB subscale | 17.6 (6.12) | 17.8 (5.98) |  |
  End of Treatment, FWB subscale: number analyzed (Participants) | 184 | 182 | 0 | 0
  End of Treatment, FWB subscale | 16.5 (6.24) | 16.3 (6.19) |  |
  Baseline, FACT-LymS: number analyzed (Participants) | 260 | 264 | 0 | 0
  Baseline, FACT-LymS | 47.7 (8.87) | 47.7 (7.88) |  |
  End of Treatment, FACT-LymS: number analyzed (Participants) | 183 | 183 | 0 | 0
  End of Treatment, FACT-LymS | 48.0 (9.41) | 48.0 (8.98) |  |
  Baseline, FACT-Lymphoma TOI: number analyzed (Participants) | 258 | 262 | 0 | 0
  Baseline, FACT-Lymphoma TOI | 89.3 (16.07) | 89.8 (15.51) |  |
  End of Treatment, FACT-Lymphoma TOI: number analyzed (Participants) | 183 | 180 | 0 | 0
  End of Treatment, FACT-Lymphoma TOI | 88.0 (17.80) | 87.3 (18.59) |  |
  Baseline, FACT-G Total Score: number analyzed (Participants) | 259 | 262 | 0 | 0
  Baseline, FACT-G Total Score | 80.7 (15.04) | 80.9 (15.08) |  |
  End of Treatment, FACT-G Total Score: number analyzed (Participants) | 182 | 178 | 0 | 0
  End of Treatment, FACT-G Total Score | 78.3 (16.63) | 77.3 (17.02) |  |
  Baseline, FACT-Lymphoma Total Score: number analyzed (Participants) | 258 | 261 | 0 | 0
  Baseline, FACT-Lymphoma Total Score | 128.4 (21.81) | 128.6 (21.27) |  |
  End of Treatment, FACT-Lymphoma Total Score: number analyzed (Participants) | 181 | 178 | 0 | 0
  End of Treatment, FACT-Lymphoma Total Score | 126.1 (24.39) | 125.2 (24.65) |  |

36. Secondary Outcome: Overall Population: FACT-Lym Scores at Baseline and End of Treatment
Description: as for outcome 35
Time Frame: up to approximately 34 months
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | FL and MZL: Tafasitamab + Rituximab + Lenalidomide | FL and MZL: Placebo + Rituximab + Lenalidomide
Number analyzed (Participants) | 326 | 328
scores on a scale
  Baseline, PWB subscale: number analyzed (Participants) | 308 | 311
  Baseline, PWB subscale | 23.8 (4.41) | 24.1 (4.20)
  End of Treatment, PWB subscale: number analyzed (Participants) | 225 | 225
  End of Treatment, PWB subscale | 23.6 (4.71) | 23.2 (5.21)
  Baseline, SWB subscale: number analyzed (Participants) | 310 | 312
  Baseline, SWB subscale | 20.8 (5.82) | 20.2 (6.06)
  End of Treatment, SWB subscale: number analyzed (Participants) | 223 | 223
  End of Treatment, SWB subscale | 20.2 (5.89) | 19.8 (5.34)
  Baseline, EWB subscale: number analyzed (Participants) | 311 | 313
  Baseline, EWB subscale | 18.2 (4.20) | 18.1 (4.12)
  End of Treatment, EWB subscale: number analyzed (Participants) | 225 | 225
  End of Treatment, EWB subscale | 18.7 (4.31) | 18.1 (4.67)
  Baseline, FWB subscale: number analyzed (Participants) | 311 | 312
  Baseline, FWB subscale | 17.3 (6.19) | 17.3 (6.08)
  End of Treatment, FWB subscale: number analyzed (Participants) | 225 | 224
  End of Treatment, FWB subscale | 16.8 (6.29) | 16.2 (6.22)
  Baseline, FACT-LymS: number analyzed (Participants) | 310 | 312
  Baseline, FACT-LymS | 47.4 (8.91) | 47.6 (7.98)
  End of Treatment, FACT-LymS: number analyzed (Participants) | 224 | 225
  End of Treatment, FACT-LymS | 48.7 (9.17) | 48.2 (8.71)
  Baseline, FACT-Lymphoma TOI: number analyzed (Participants) | 307 | 309
  Baseline, FACT-Lymphoma TOI | 88.7 (16.40) | 89.0 (15.72)
  End of Treatment, FACT-Lymphoma TOI: number analyzed (Participants) | 224 | 222
  End of Treatment, FACT-Lymphoma TOI | 89.0 (17.74) | 87.4 (18.14)
  Baseline, FACT-G Total Score: number analyzed (Participants) | 308 | 309
  Baseline, FACT-G Total Score | 80.2 (15.39) | 79.7 (15.43)
  End of Treatment, FACT-G Total Score: number analyzed (Participants) | 223 | 220
  End of Treatment, FACT-G Total Score | 79.2 (16.65) | 77.1 (16.80)
  Baseline, FACT-Lymphoma Total Score: number analyzed (Participants) | 307 | 308
  Baseline, FACT-Lymphoma Total Score | 127.7 (22.18) | 127.3 (21.57)
  End of Treatment, FACT-Lymphoma Total Score: number analyzed (Participants) | 222 | 220
  End of Treatment, FACT-Lymphoma Total Score | 127.8 (24.26) | 125.2 (24.18)

ADVERSE EVENTS:
Time Frame: from signing of the Informed Consent Form to up to 90 days post-treatment (up to approximately 3 years)
Description: As pre-specified in the Statistical Analysis Plan, the MZL population was considered as a subpopulation of interest, not a main analysis population. The FL and MZL populations were combined for analysis into the Overall population, which was a main analysis population. Safety was not expected to be different between each histological subtype (FL versus MZL).
Groups:
- Tafasitamab + Rituximab + Lenalidomide: Participants with follicular lymphoma (FL) or marginal zone lymphoma (MZL) were randomized to receive tafasitamab 12 milligrams per kilogram (mg/kg) intravenously (IV), administered on Days 1, 8, 15, and 22 of Cycles 1 to 3 and on Days 1 and 15 of Cycles 4 to 12. Participants also received oral lenalidomide (including generics) 20 mg once daily (QD), administered at approximately the same time every day on Days 1 to 21 of Cycles 1 to 12, and rituximab (including biosimilars) 375 mg/meters squared (m^2) IV, administered on Days 1, 8, 15, and 22 of Cycle 1 and on Day 1 of Cycles 2 to 5. A treatment cycle was defined as 28 calendar days.
- Placebo + Rituximab + Lenalidomide: Participants with FL or MZL were randomized to receive placebo 0.9% saline solution IV, administered on Days 1, 8, 15, and 22 of Cycles 1 to 3 and on Days 1 and 15 of Cycles 4 to 12. Participants also received oral lenalidomide (including generics) 20 mg QD, administered at approximately the same time every day on Days 1 to 21 of Cycles 1 to 12, and rituximab (including biosimilars) 375 mg/m^2 IV, administered on Days 1, 8, 15, and 22 of Cycle 1 and on Day 1 of Cycles 2 to 5. A treatment cycle was defined as 28 calendar days.
- Total: Total
Arm/Group | Tafasitamab + Rituximab + Lenalidomide | Placebo + Rituximab + Lenalidomide | Total
All-Cause Mortality (participants affected / at risk) | 22/327 | 24/325 | 46/652
Serious Adverse Events (participants affected / at risk) | 125/327 | 110/325 | 235/652
Other Adverse Events (participants affected / at risk) | 318/327 | 315/325 | 633/652
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tafasitamab + Rituximab + Lenalidomide (N=327) | Placebo + Rituximab + Lenalidomide (N=325) | Total (N=652)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 5 (5) | 5 (5)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 9 (9) | 6 (6) | 15 (15)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 3 (3)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 5 (5)
Anal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 21 (27) | 8 (9) | 29 (36)
COVID-19 pneumonia (Infections and infestations) | 17 (19) | 7 (8) | 24 (27)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Carcinoid tumour in the large intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2) | 4 (4)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2) | 3 (3)
Device related infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Device related thrombosis (General disorders) | 0 (0) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (4)
Embolism (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (10) | 10 (11) | 19 (21)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Haemophilus bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatosplenomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperthermia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Infective exacerbation of asthma (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (2) | 0 (0) | 1 (2)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 2 (2) | 3 (4)
Lymphatic fistula (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2) | 2 (2)
Moraxella infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Myopericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (5) | 3 (4) | 5 (9)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Norovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (4)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 25 (33) | 15 (18) | 40 (51)
Pneumonia adenoviral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia moraxella (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Prostatic abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pseudomonal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 6 (7) | 11 (12) | 17 (19)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 6 (6)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 4 (4) | 5 (5) | 9 (9)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Serum sickness (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 4 (4)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 4 (4)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Varicella zoster pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tafasitamab + Rituximab + Lenalidomide (N=327) | Placebo + Rituximab + Lenalidomide (N=325) | Total (N=652)
Abdominal pain (Gastrointestinal disorders) | 25 (33) | 28 (30) | 53 (63)
Alanine aminotransferase increased (Investigations) | 19 (28) | 23 (36) | 42 (64)
Anaemia (Blood and lymphatic system disorders) | 53 (97) | 46 (73) | 99 (170)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (25) | 27 (36) | 51 (61)
Asthenia (General disorders) | 44 (58) | 35 (48) | 79 (106)
Back pain (Musculoskeletal and connective tissue disorders) | 32 (41) | 18 (21) | 50 (62)
Bronchitis (Infections and infestations) | 17 (21) | 14 (14) | 31 (35)
COVID-19 (Infections and infestations) | 86 (98) | 72 (81) | 158 (179)
Chills (General disorders) | 14 (14) | 17 (18) | 31 (32)
Constipation (Gastrointestinal disorders) | 90 (110) | 81 (100) | 171 (210)
Cough (Respiratory, thoracic and mediastinal disorders) | 62 (81) | 55 (69) | 117 (150)
Decreased appetite (Metabolism and nutrition disorders) | 36 (39) | 30 (32) | 66 (71)
Diarrhoea (Gastrointestinal disorders) | 123 (219) | 101 (162) | 224 (381)
Dizziness (Nervous system disorders) | 26 (34) | 23 (28) | 49 (62)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 (26) | 30 (32) | 52 (58)
Fatigue (General disorders) | 67 (80) | 53 (64) | 120 (144)
Headache (Nervous system disorders) | 34 (47) | 25 (30) | 59 (77)
Hypokalaemia (Metabolism and nutrition disorders) | 27 (44) | 41 (60) | 68 (104)
Hypotension (Vascular disorders) | 20 (22) | 14 (16) | 34 (38)
Infusion related reaction (Injury, poisoning and procedural complications) | 52 (58) | 49 (61) | 101 (119)
Insomnia (Psychiatric disorders) | 25 (25) | 23 (23) | 48 (48)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 53 (68) | 57 (64) | 110 (132)
Myalgia (Musculoskeletal and connective tissue disorders) | 20 (21) | 15 (20) | 35 (41)
Nasopharyngitis (Infections and infestations) | 19 (22) | 21 (22) | 40 (44)
Nausea (Gastrointestinal disorders) | 59 (76) | 47 (58) | 106 (134)
Neutropenia (Blood and lymphatic system disorders) | 164 (470) | 154 (388) | 318 (858)
Neutrophil count decreased (Investigations) | 24 (65) | 23 (60) | 47 (125)
Oedema peripheral (General disorders) | 25 (27) | 44 (45) | 69 (72)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 29 (37) | 14 (15) | 43 (52)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 (28) | 11 (12) | 34 (40)
Pruritus (Skin and subcutaneous tissue disorders) | 51 (70) | 38 (49) | 89 (119)
Pyrexia (General disorders) | 60 (85) | 49 (63) | 109 (148)
Rash (Skin and subcutaneous tissue disorders) | 72 (103) | 70 (115) | 142 (218)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 (22) | 16 (26) | 34 (48)
Respiratory tract infection (Infections and infestations) | 21 (33) | 26 (32) | 47 (65)
Thrombocytopenia (Blood and lymphatic system disorders) | 48 (121) | 59 (91) | 107 (212)
Upper respiratory tract infection (Infections and infestations) | 28 (37) | 36 (40) | 64 (77)
Urinary tract infection (Infections and infestations) | 26 (34) | 21 (27) | 47 (61)
Vomiting (Gastrointestinal disorders) | 24 (28) | 16 (20) | 40 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT04680052/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT04680052/SAP_001.pdf